CLINICAL TRIAL: NCT03422419
Title: An Investigator-initiated, Multicentre, Randomized, Trial Comparing Anticoagulation Alone Versus Transjugular Intrahepatic Portosystemic Shunt (TIPS) and Anticoagulation in Patients With Recent Obstructive Portal Vein Thrombosis
Brief Title: TIPS or Anticoagulation in Portal Vein Thrombosis
Acronym: PROGRESS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IICT2017_PROGRESS
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Thrombosis Portal Vein
MeSH Terms: interventions — Heparin; Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIPS+Anticoagulation (Experimental)
  Interventions: Drug: Heparin; Device: TIPS
- Anticoagulation (Active Comparator)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — The choice of the anticoagulant medication in terms of duration and dose will be determined by the treating physician.
Device: TIPS — transjugular intrahepatic portosystemic shunt deployment
  Arms: TIPS+Anticoagulation

SUMMARY:
The PROGRESS is an investigator-initiated, multicentre, randomized, trial comparing anticoagulation, which is the currently most frequently used treatment, alone, versus transjugular intrahepatic portosystemic shunt (TIPS) combined with anticoagulation, in patients presenting with recent obstructive portal vein thrombosis (ROPVT). The rationale of this study is to significantly increase the proportion of patients that achieve a complete or partial recanalization of the portal vein. The intervention of this study consists in TIPS deployment and catheter based clot removal in addition to anticoagulation. The investigators retain that this intervention will increase the proportion of patients with an open portal vein from 38% with anticoagulation alone to 83% with anticoagulation and TIPS after 6 months. Both anticoagulant therapy and clot removal/TIPS are treatments that are currently available and accepted indications for the treatment of ROPVT. Anticoagulation will be performed with unfractioned heparin or low molecular weight heparin initially and with vitamin K antagonists in the long term. The investigators plan to collect blood for biobanking at the time of inclusion and after 6 months. Blood samples for a biobank will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Recent complete thrombosis of the extrahepatic portal vein either with or without the involvement of intrahepatic branches and with or without involvement of splenic vein and superior mesenteric vein
2. Written informed consent

Exclusion Criteria:

1. Malignant Portal Vein thrombosis (neoplastic invasion)
2. Intraabdominal malignancy
3. Chronic diseases limiting life expectancy in the short term (6 months)
4. Liver transplantation
5. Unwillingness to participate
6. Contraindications to TIPS (including past or present hepatic encephalopathy Grade ≥2)
7. Child-Pugh-Turcotte score 11 or more points in patients with advanced chronic liver disease-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete recanalization of the portal vein". | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Gottardi, Prof. Dr. med, Principal Investigator — Insel Gruppe AG, University Hospital Bern

IPD SHARING:
Plan to Share IPD: Undecided